CLINICAL TRIAL: NCT03305328
Title: Assessing the Clinical Utility of tACS in the Treatment of Anxious Arousal and Sensory Sensitivity
Brief Title: Assessing the Clinical Utility of tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Wen Li, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.20700
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Anxiety Disorders and Symptoms; Sensory Disorders; Hypervigilance; Post Traumatic Stress Disorder
Keywords: Oscillations; Non-invasive Brain Stimulation; Transcranial Alternating Current Stimulation
MeSH Terms: conditions — Anxiety Disorders; Sensation Disorders; Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an Active or Sham Control group. The Active group received the 30 minutes of alpha-tACS for four consecutive days, whereas the Sham Control group received Sham (no) stimulation.
Who Masked: Participant
Masking Description: Participants were unaware of the presence of a Sham condition. Therefore, all participants believed they received the Active stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Participants within the Active condition receive 30 minutes of alpha-frequency Transcranial Alternating Current Stimulation (tACS) stimulation for four consecutive days. Participants are stimulated at their baseline peak alpha frequency, or the frequency at which they exhibit maximal power within the 8 to 12 Hz range. Stimulation was administered over occipitoparietal sites, where tACS current models showed maximal effect over the dorsal extrastriate.
  Interventions: Device: Transcranial Alternating Current Stimulation
- Sham Control (Sham Comparator): Participants within the Sham condition receive 30 minutes of sham Transcranial Alternating Current Stimulation for four consecutive days, during which no current was passed. To control for awareness of the Sham stimulation, all Sham control participants receive a brief, 10 second pulse of random noise stimulation at the beginning and end of the 30 minutes.
  Interventions: Device: Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Transcranial Alternating Current Stimulation passes a weak, 2 mA sinusoidal current through the scalp to the cortex at a specified frequency. Previous evidence suggests this exogenous sinusoidal stimulation interacts with the endogenous, cortical sinusoidal oscillatory activity, resulting in modulations of cortical oscillations. The intervention is non-invasive and virtually painless with no lasting adverse side-effects.

SUMMARY:
The present study seeks to evaluate the clinical utility of repeated transcranial alternating current stimulation (tACS) by assessing long-term, lasting changes in oscillatory activity and subsequent changes in related behavioral processes of anxious arousal and sensory sensitivity. To date, only transient effects of tACS have been reported, lasting no longer than 30 to 70 minutes. In order to be truly impactful within a clinical setting, however, evidence for long-term effects of tACS is needed.

DETAILED DESCRIPTION:
Recent years have witnessed increasing recognition of "oscillopathies", neuropsychiatric disorders characterized by aberrations in the neural oscillations that orchestrate various mental activities. Transcranial alternating current stimulation (tACS) provides an effective way to directly modulate these oscillations in a non-invasive and frequency-specific manner, offering groundbreaking insights into the workings of the brain and, importantly, the development of novel treatments for these oscillopathies. However, evidence is lacking for the ability of tACS to induce long-term neural plasticity and lasting behavioral changes, which is critical for establishing the clinical utility of this novel intervention.

Here, we are administering 30 minutes of alpha-frequency tACS over occipitoparietal sites for four consecutive days to evaluate both transient and long-term changes in alpha oscillatory power and long-range, directed oscillatory connectivity. As both anxious arousal and sensory sensitivity are highly related to alpha oscillations, as well as numerous neuropsychiatric disorders, changes in these behavioral outcomes were subsequently evaluated to assess clinically-relevant outcomes of the repeated tACS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed

Exclusion Criteria:

* History of severe neurological disorder or traumatic brain injury
* Psychotropic medication use
* Metal plates/implants in head
* Pregnancy
* Implanted medical devices (e.x. pacemaker)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Immediate and lasting changes in alpha oscillatory power and directed, long-range cortico-cortical connectivity. | Immediately before, immediately after, and 30 minutes after stimulation on the first day. Immediately before (24 hours after most recent stimulation), immediately after, and 30 minutes after stimulation on the final (fourth) day.
  Occipitoparietal alpha power and long-range, directed oscillatory connectivity within the alpha frequency will be assessed from 2 minutes of eyes-open, resting-state electroencephalogram (EEG) activity. Oscillatory power will be estimated using the multitaper spectral estimation technique, averaging over the alpha frequency bin of 8-12 Hz. Directed connectivity will be assessed using spectral Granger causality within the 8-12 Hz range. Specifically, long-range, posterior-frontal connectivity with be assessed.

SECONDARY OUTCOMES:
Immediate and lasting reductions in anxious arousal | Immediately before, immediately after, 30 minutes after stimulation on the first and final day. Immediately before (24 hours after most recent stimulation) and immediately after stimulation on the second and third days.
  Self-report ratings of subjective units of anxious arousal are acquired using a visual analog scale, ranging from 0 (not at all anxiously aroused) to 100 (extremely anxiously aroused).
Immediate and lasting changes in affective perception of sensory stimuli | Immediately before, immediately after, and 30 minutes after stimulation on the first day. Immediately before (24 hours after most recent stimulation), immediately after, and 30 minutes after stimulation on the final (fourth) day.
  Pleasantness ratings of neutral and negative olfactory and auditory stimuli are acquired on a visual analog scale, ranging from 0 (extremely unpleasant) to 100 (extremely pleasant). Auditory stimuli consist of a simple tone (neutral) and scream (negative) at three different intensities (quiet, medium, and loud), each presented once for 2 seconds through headphones. Olfactory stimuli consist of a neutral odor (acetophenone) and negative odor (burning rubber), diluted in mineral oil for three different intensities (weak, medium, strong). Approximately 3 mL of each odor are presented in 30 mL amber bottles, upon which participants are asked to take one steady sniff.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, PhD, Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: Undecided